CLINICAL TRIAL: NCT00294346
Title: A Phase 2, Double-Blind, Placebo-Controlled Trial to Investigate the Safety and Efficacy of AV608 in Subjects With Social Anxiety Disorder
Brief Title: Safety and Efficacy Study of AV608 in Subjects With Social Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avera Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AV608-105
Record Dates: First submitted 2006-02-17; First posted 2006-02-22 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2008-02

CONDITIONS: Social Phobia
Keywords: Social Anxiety Disorder; Social Phobia
MeSH Terms: conditions — Phobia, Social

INTERVENTIONS:
Drug: AV608

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of an investigational drug (AV608) when used in subjects who have Social Anxiety Disorder. AV608 is an NK-1 receptor antagonist that exhibits central nervous system activity after oral administration. The study will compare AV608 to placebo (a medically inactive substance) to see if AV608 helps the symptoms of Social Anxiety Disorder. Eligible subjects will be assigned by chance to take either AV608 or placebo for 12 weeks. During the study, subjects will be asked about their overall health and mood and their Social Anxiety Disorder.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female, 18 - 65 years of age (inclusive).
2. The subject meets current DSM-IV-TR (American Psychiatric Association, 2000) criteria for Social Phobia (300.23), generalized subtype, as confirmed by the Mini-International Neuropsychiatric Interview at Screening (Visit 1).
3. The subject has had symptoms of SAD (Social Phobia) present for at least 6 months prior to Screening (Visit 1).
4. The subject has a total score ≥ 60 on the LSAS at both Screening (Visit 1) and Baseline (Visit 2).
5. The subject has a score ≥ 4 on the Clinical Global Impression - Severity (CGI-S) scale at both Screening (Visit 1) and Baseline (Visit 2).
6. The subject has a score ≤ 15 on the 17-item Hamilton Rating Scale for Depression (HAM-D) at Screening
7. The subject, if female and of child-bearing potential (not 2 years post-menopausal or surgically sterilized), must have a negative serum pregnancy test at Screening (Visit 1) and be willing to avoid pregnancy and practice adequate birth control from the time of study enrollment until 30 days after the last dose of study medication. Adequate methods of birth control are: oral contraception, intrauterine device, implantable contraceptive device, depot contraceptive, or a barrier method plus spermicide. Additional serum pregnancy tests will be administered at Visit 6, Visit 8, and Visit 9.
8. The subject, if engaged in ongoing psychotherapy for SAD or any other mental health condition, must have been attending therapy regularly for at least 3 months prior to Screening (Visit 1) and must agree to continue the same type and frequency of psychotherapy throughout the course of the study.
9. The subject agrees to refrain from blood donation during the course of the study.
10. The subject has written and oral fluency in English or Spanish.
11. The subject is willing to participate in the study, as evidenced by a signed and dated written Informed Consent Form (ICF).

Exclusion Criteria:

1. The subject has a decrease >15 points on the LSAS total score between Screening (Visit 1) and Baseline (Visit 2).
2. The subject has a clinically significant abnormality or clinically significant unstable medical condition as indicated by medical history, physical examination, ECG results, clinical laboratory testing, or the investigator's judgment at Screening (Visit 1) or Baseline (Visit 2).
3. The subject has a QTc interval of 450 msec or greater at Screening (Visit 1) if male or a QTc interval of 470 msec or greater at Screening (Visit 1) if female.
4. The subject has current hypothyroidism or hyperthyroidism or laboratory findings consistent with thyroid dysfunction. Subjects who are being treated for thyroid disorder are eligible if they have been on stable doses of thyroid hormone for at least 6 months and are currently euthyroid.
5. The subject has any history of schizophrenia or other psychotic disorder, bipolar disorder, post-traumatic stress disorder, borderline personality disorder, or antisocial personality disorder.
6. The subject has a history within the previous 5 years of obsessive-compulsive disorder or an eating disorder.
7. The subject exhibits evidence of a clinically predominant DSM-IV-TR Axis I or II disorder other than Social Phobia or Avoidant Personality Disorder within the 6 months prior to Screening (Visit 1).
8. The subject, in the opinion of the investigator, presents a significant risk of doing harm to himself, herself, or others.
9. The subject has met DSM-IV-TR criteria for alcohol or substance dependence (other than nicotine or caffeine dependence) within 6 months of Screening (Visit 1).
10. The subject has met DSM-IV-TR criteria substance abuse (other than alcohol, nicotine or caffeine abuse) within 3 months of Screening (Visit 1).
11. The subject tests positive on the urine drug screen conducted at Screening (Visit 1) for illicit drugs, including opiates, barbiturates, amphetamines, cocaine, and phencyclidine.
12. The subject is a pregnant or lactating female.
13. The subject has previously participated in a clinical trial for AV608 (previously identified as NKP608 and CGP608).
14. The subject has used any prohibited medications, or has any anticipated need or intended use of these medications during the study, including:

    * Depot injection of an antipsychotic medication within 3 months prior to Baseline (Visit 2) or use of any other antipsychotic or mood stabilizing medication within 30 days prior to Baseline (Visit 2)
    * Fluoxetine within 30 days prior to Baseline (Visit 2) or any other antidepressant medication within 14 days prior to Baseline (Visit 2)
    * Any anxiolytic or sedative-hypnotic medication within 14 days prior to Baseline (Visit 2), with the exception of eszopiclone, ramelteon, zaleplon, or zolpidem if used for sleep
    * Any other psychotropic drug or substance (prescription or over-the-counter) within 7 days prior to Baseline (Visit 2), including St. John's wort, gingko biloba, chromium picolinate, kava-kava, melatonin, DHEA, diphenhydramine, ephedra, or hydroxyzine
    * Any use of pimozide, terfenadine, astemizole, or cisapride during the study
15. The subject has used any investigational drugs, products, or devices in the 3 months prior to Screening (Visit 1).
16. The subject is a member of the investigative site staff or an immediate family member.
17. The subject has any other condition that the investigator believes would jeopardize the safety or rights of the subject or would render the subject unable to comply with the trial protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2006-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Birmingham Research Group, Inc., Birmingham, Alabama
  - Pivotal Research Centers, Mesa, Arizona
  - Southwestern Research, Inc., Beverly Hills, California
  - Affiliated Research Institute, San Diego, California
  - CNS Healthcare, Jacksonville, Florida
  - Comprehensive Neuroscience, Inc., St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - DuPont Clinical Research, Inc., Rockville, Maryland
  - Capital Clinical Research Associates, Rockville, Maryland
  - Medical Research Network, LLC, New York, New York
  - Hartford Research, Cincinnatti, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Claghorn-Lesem Research Clinic, LLP, Bellaire, Texas
  - Croft Group Research Center, San Antonio, Texas